CLINICAL TRIAL: NCT07342764
Title: A Three-Arm Open-Label Pragmatic Trial Comparing Dapagliflozin, Metformin, and Lifestyle Modification for Antipsychotic-Induced Weight Gain
Brief Title: Comparative Effectiveness of Dapagliflozin, Metformin, and Lifestyle Modification for Antipsychotic-Induced Weight Gain: An Open-Label Pragmatic Trial
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Principal Investigator, Mohammed Al Alawi MD PhD MRCPsych ARABpsych OMSBpsych, Consultant and Assistant Professor, Sultan Qaboos University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIWG2025
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Antipsychotic-induced Weight Gain (AIWG); Antipsychotic-induced Weight Gain; Schizophrenia Spectrum and Other Psychotic Disorders
Keywords: Dapagliflozin; Metformin; Antipsychotic-induced weight gain; Schizophrenia; Psychotic disorders; Randomized controlled trial; Weight management; Metabolic side effects; Lifestyle intervention; SGLT2 inhibitor
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders; Schizophrenia; Psychotic Disorders | interventions — Metformin; dapagliflozin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A (Active Comparator)
  Interventions: Drug: Metformin (1000 mg Twice a day); Other: Lifestyle Modification Program
- Arm B (Experimental)
  Interventions: Drug: Dapagliflozin 10 mg; Other: Lifestyle Modification Program
- Arm C (Other): Control
  Interventions: Other: Lifestyle Modification Program

INTERVENTIONS:
Drug: Metformin (1000 mg Twice a day) — Metformin tablets starting at 500 mg twice daily and increased to 1000 mg twice daily as tolerated, taken with meals for 26 weeks.
  Arms: Arm A
Drug: Dapagliflozin 10 mg — Dapagliflozin 10 mg tablet taken once daily for 26 weeks. It increases glucose excretion through urine and may lower weight.
  Arms: Arm B
Other: Lifestyle Modification Program — Participants receive a structured lifestyle program, including dietary counseling, physical-activity planning, and behavioral support at scheduled visits (weeks 0, 4, 12, and 26).

SUMMARY:
Clinical trial:

The goal of this clinical trial is to learn if dapagliflozin can help reduce weight gain caused by antipsychotic medications in people with schizophrenia and related disorders. It will also assess the safety of dapagliflozin.

* The main questions it aims to answer are:

  * Does dapagliflozin lower body weight compared to metformin or lifestyle changes alone?
  * Does it improve blood sugar, cholesterol, and overall health?
* Researchers will compare three groups:

  * Dapagliflozin plus lifestyle changes
  * Metformin plus lifestyle changes
  * Lifestyle changes alone
* Participants will:

  * Take the assigned medication daily for 26 weeks (or follow lifestyle guidance only)
  * Attend clinic visits at weeks 0, 4, 12, and 26 for measurements and blood tests
  * Receive phone calls for follow-up and side effect checks

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn whether a medication called dapagliflozin can help reduce weight gain caused by antipsychotic medicines. These medicines are important for treating conditions like schizophrenia, but they often lead to weight gain and other metabolic problems such as changes in blood sugar and cholesterol. This can make it harder for people to continue their treatment.

3 Researchers will compare three different approaches to see which works best to help with antipsychotic-related weight gain:

* Metformin plus lifestyle changes (diet and exercise guidance)
* Dapagliflozin plus lifestyle changes
* Lifestyle changes alone

  # The main question the study aims to answer is:
* Does dapagliflozin help people lose more weight or prevent further weight gain compared to lifestyle changes alone or metformin?

  # Other questions include:
* How do these approaches affect blood sugar, cholesterol, and overall health?
* How well do participants tolerate dapagliflozin compared to metformin?
* Do these treatments improve quality of life and treatment satisfaction?

  * Study Design This is a 26-week randomized controlled trial taking place at Sultan Qaboos University Hospital in Muscat, Oman.

Participants will be randomly assigned to one of the three groups above. Neither the participants nor their doctors will be blinded, but the researchers who measure results and analyze the data will not know which group participants are in, to keep the results fair.

Who Can Take Part

People aged 16 years or older who:

* Have a schizophrenia-spectrum disorder (as defined in DSM-5)
* Are taking one antipsychotic medicine and have been stable for at least 3 months
* Have gained 7% or more of their body weight since starting the medication, or have a BMI over 25 kg/m²

People cannot join if they:

* Have diabetes, kidney, or liver disease
* Are pregnant or breastfeeding
* Have recently used weight-loss medications
* Have unstable mental illness or substance use that affects study participation

What Participants Will Do All participants will receive lifestyle guidance, including diet, exercise, and behavioral support.

In addition:

* One group will take metformin tablets twice daily
* One group will take dapagliflozin once daily
* One group will make lifestyle changes only

Participants will:

* Visit the clinic at the start, and again at weeks 4, 12, and 26
* Receive phone calls at weeks 2, 8, and 18 to check on progress and side effects
* Have blood tests and measurements (weight, waist, glucose, cholesterol)
* Fill out questionnaires about physical activity, mood, and quality of life

What the Study Will Measure

* Main outcome: Change in body weight after 26 weeks
* Other outcomes:

BMI and waist circumference Blood sugar, insulin, and cholesterol levels Percentage of people losing 5% or more of their weight Psychiatric symptom scores and quality of life Any side effects or treatment satisfaction

Why This Research Matters Many people who take antipsychotics struggle with weight gain, which can harm their health and make them stop treatment. Dapagliflozin is already used for diabetes and helps the body remove extra sugar through urine, which may also help reduce weight gain. However, no study has yet tested dapagliflozin specifically for antipsychotic-induced weight gain.

This research could identify a new, safe, and effective way to manage this problem, helping people stay healthy and continue their psychiatric treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years or older.
* Diagnosis of a schizophrenia spectrum or other psychotic disorder according to DSM-5 (excluding substance/medication-induced or medical-condition-related psychoses, catatonia due to another disorder, or unspecified catatonia).
* On stable antipsychotic monotherapy for at least 3 months before enrollment.
* Evidence of antipsychotic-induced weight gain, defined as:

  * ≥7% increase in body weight from pre-treatment baseline, or
  * Body Mass Index (BMI) >25 kg/m² with documented antipsychotic-related weight gain.
* Stable psychiatric symptoms, judged clinically able to give informed consent and participate in the study.

Exclusion Criteria:

* Diabetes mellitus (type 1 or type 2).
* Renal impairment (estimated glomerular filtration rate <45 mL/min/1.73 m²), hepatic disease, or other serious medical illness.
* Pregnancy or breastfeeding.
* Use of weight-loss medications or programs within the past 3 months.
* Known hypersensitivity to metformin or dapagliflozin.
* Unstable psychiatric condition or active substance use disorder likely to interfere with adherence or follow-up.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Body Weight | 26 weeks
  Percentage change in body weight from baseline to week 26, measured using a calibrated digital scale. This assesses whether dapagliflozin or metformin combined with lifestyle modification reduces antipsychotic-induced weight gain compared to lifestyle modification alone.

SECONDARY OUTCOMES:
Change in Body Mass Index (BMI) | 26 weeks
  Change in BMI (kg/m²) from baseline to week 26 to evaluate overall body composition changes associated with each intervention.
Change in Waist Circumference | 26 weeks
  Change in waist circumference (measured at the midpoint between the lowest rib and iliac crest) from baseline to week 26, assessing central fat distribution.
Change in Fasting Plasma Glucose | 26 weeks
  Difference in fasting plasma glucose levels from baseline to week 26, reflecting glucose metabolism and glycemic control.
Change in Glycated Hemoglobin (HbA1c) | 26 weeks
  Change in HbA1c (%) from baseline to week 26, assessing long-term glucose regulation.
Change in Lipid Profile | 26 weeks
  Change in total cholesterol, LDL, HDL, and triglycerides from baseline to week 26, evaluating metabolic health and cardiovascular risk.
Change in Psychiatric Symptom Severity (PANSS or BPRS) | 26 weeks
  Change in Positive and Negative Syndrome Scale (PANSS) or Brief Psychiatric Rating Scale (BPRS) total scores to evaluate the impact of interventions on psychiatric stability.
Incidence of Adverse Events | 26 weeks
  Frequency and type of treatment-emergent adverse events recorded throughout the study period to evaluate safety and tolerability of each intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Al Alawi, MD, PhD, Study Chair — Sultan Qaboos University
Locations (1):
- SQU, Muscat, Oman

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferreira-Hermosillo A, Molina-Ayala MA, Molina-Guerrero D, Garrido-Mendoza AP, Ramirez-Renteria C, Mendoza-Zubieta V, Espinosa E, Mercado M. Efficacy of the treatment with dapagliflozin and metformin compared to metformin monotherapy for weight loss in patients with class III obesity: a randomized controlled trial. Trials. 2020 Feb 14;21(1):186. doi: 10.1186/s13063-020-4121-x. PMID 32059692
- [Background] Bolinder J, Ljunggren O, Johansson L, Wilding J, Langkilde AM, Sjostrom CD, Sugg J, Parikh S. Dapagliflozin maintains glycaemic control while reducing weight and body fat mass over 2 years in patients with type 2 diabetes mellitus inadequately controlled on metformin. Diabetes Obes Metab. 2014 Feb;16(2):159-69. doi: 10.1111/dom.12189. Epub 2013 Aug 29. PMID 23906445
- [Background] Bolinder J, Ljunggren O, Kullberg J, Johansson L, Wilding J, Langkilde AM, Sugg J, Parikh S. Effects of dapagliflozin on body weight, total fat mass, and regional adipose tissue distribution in patients with type 2 diabetes mellitus with inadequate glycemic control on metformin. J Clin Endocrinol Metab. 2012 Mar;97(3):1020-31. doi: 10.1210/jc.2011-2260. Epub 2012 Jan 11. PMID 22238392
- [Background] Mansuri Z, Makani R, Trivedi C, Adnan M, Vadukapuram R, Rafael J, Lodhi A, Reddy A. The role of metformin in treatment of weight gain associated with atypical antipsychotic treatment in children and adolescents: A systematic review and meta-analysis of randomized controlled trials. Front Psychiatry. 2022 Nov 15;13:933570. doi: 10.3389/fpsyt.2022.933570. eCollection 2022. PMID 36458118
- [Background] Hegde NC, Mishra A, Maiti R, Mishra BR, Mohapatra D, Srinivasan A. Pharmacological interventions for antipsychotic-induced weight gain in schizophrenia: A network meta-analysis. Gen Hosp Psychiatry. 2024 Sep-Oct;90:12-21. doi: 10.1016/j.genhosppsych.2024.06.003. Epub 2024 Jun 11. PMID 38878592
- [Background] de Silva VA, Suraweera C, Ratnatunga SS, Dayabandara M, Wanniarachchi N, Hanwella R. Metformin in prevention and treatment of antipsychotic induced weight gain: a systematic review and meta-analysis. BMC Psychiatry. 2016 Oct 3;16(1):341. doi: 10.1186/s12888-016-1049-5. PMID 27716110
- [Background] Dayabandara M, Hanwella R, Ratnatunga S, Seneviratne S, Suraweera C, de Silva VA. Antipsychotic-associated weight gain: management strategies and impact on treatment adherence. Neuropsychiatr Dis Treat. 2017 Aug 22;13:2231-2241. doi: 10.2147/NDT.S113099. eCollection 2017. PMID 28883731
- [Background] Musil R, Obermeier M, Russ P, Hamerle M. Weight gain and antipsychotics: a drug safety review. Expert Opin Drug Saf. 2015 Jan;14(1):73-96. doi: 10.1517/14740338.2015.974549. Epub 2014 Nov 15. PMID 25400109
- [Background] Barton BB, Segger F, Fischer K, Obermeier M, Musil R. Update on weight-gain caused by antipsychotics: a systematic review and meta-analysis. Expert Opin Drug Saf. 2020 Mar;19(3):295-314. doi: 10.1080/14740338.2020.1713091. Epub 2020 Mar 12. PMID 31952459